CLINICAL TRIAL: NCT02332746
Title: Novel Exploration of Temporal Relationships Between Self-worth and Physical Activity in Middle-aged Women
Brief Title: Exploring Temporal Relationships Between Self-worth and Physical Activity Middle-aged Women
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Other Study IDs: 1308009564
Record Dates: First submitted 2014-12-18; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Self Esteem; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Middle-aged women: Middle-aged women (35-64 years)

SUMMARY:
The purpose of this study is to explore temporal relationships between self-worth and physical activity (PA) participation in middle-aged women (aged 35-64 years). We are particularly interested in the predictive role of self-worth on women's daily PA participation.

This study will include two phases: a pilot phase to test the procedures and a test phase to assess self-worth and PA. During the test phase, Women will receive text message prompts in the morning, afternoon, and evening for 28 days on their cell phones. Each prompt will include a link to an 11-item mobile Internet-based survey assessing momentary PA, self-worth, and self-efficacy. Women will also concurrently wear an activity monitor (GENEActiv) to objectively measure their activity levels throughout the study.

DETAILED DESCRIPTION:
Using ecological momentary assessment, the purpose of this study is to explore temporal relationships between self-worth and physical activity (PA) participation in middle-aged women (aged 35-64 years).

This study will occur in two phases. During an initial pilot phase ten women will be asked to test the instruments and procedures for this study. During the second phase, the test phase, 60-100 women will be asked to complete daily surveys assessing their self-worth, self-efficacy, and PA participation. The results of the pilot phase will be used to modify instruments and procedures before the test phase commences.

During the pilot phase, 10 women will be asked to participate in an initial intake appointment to sign the informed consent form, complete baseline questionnaires, receive an activity monitor, and receive instructions on completing the daily surveys and wearing the activity monitor. Women will also be asked to provide their typical daily wake times and bedtimes during this appointment to guide the sampling schedule. Ecological momentary assessment (EMA) in which women receive two or three daily prompts to complete a short survey will be used in this study. Women will be asked to answer seven questions assessing their momentary activity (1), self-efficacy (1), and self-worth (5) twice per day for one week and three times per day for one week. Five women will be assigned to each condition each week so that half of the sample receives the twice per day condition during the first week and half receives the twice per day condition during the second week of the pilot phase. Women sampled twice per day will be prompted to complete assessments 1) 15 minutes after their typical wake time reported during their intake appointment and 2) 90 minutes prior to their typical bedtime. Women sampled three times per day will be prompted one additional time during the afternoon (random time between 2:00 and 3:00pm). Women will be prompted to complete the survey via text message. A link will be provided in each text message to direct women to a mobile compatible Qualtrics survey containing seven items assessing women's current activity, self-efficacy, general self-worth, knowledge self-worth, emotional self-worth, social self-worth, and physical self-worth. At the end of the two week pilot phase, women will be asked to complete a survey to provide feedback on the sampling scheme and the usability of the mobile survey. Results of the survey will inform modifications to the test phase.

During the test phase, 60-100 women will be asked to participate in an initial intake appointment to sign the informed consent form, complete baseline questionnaires, receive an activity monitor, and receive instructions on completing the daily surveys and wearing the activity monitor. Women will be asked to answer eleven questions assessing their current activity (1), self-efficacy (1), and self-worth (9) three times per day for 28 days, depending upon the results of the pilot phase. The three-times daily sampling scheme will be adopted for the test phase. Therefore, women will receive text message prompts with a link to the mobile compatible Qualtrics survey daily in the morning, afternoon, and evening.

Current activity will be measured using an item modified from a recent EMA study by Dunton and colleagues (2012). Using a list of options, this item assesses the activity in which the participant was engaged immediately prior to receiving the prompt. One item from the Exercise Self-Efficacy Scale (McAuley, 1993) will be used to assess women's confidence in their ability to participate in daily PA on a scale of 0% to 100% - "I am able to participate in physical activity at a moderate intensity for 30+ minutes today without quitting." General self-worth will be measured using one item from the general self-worth subscale of the Adult Self-Perception Profile (Messer & Harter, 1986). Women will choose among four statements to indicate how they feel about themselves: "Which of the following statements is most true of how you feel RIGHT NOW? It is REALLY TRUE that I am dissatisfied with myself It is SORT OF TRUE that I am dissatisfied with myself It is SORT OF TRUE that I am satisfied with myself It is REALLY TRUE that I am satisfied with myself"

The Women's Physical Activity Self-Worth Inventory (WPASWI) (Huberty et al., 2013) will be used to measure knowledge, emotional, and social self-worth. Women will be asked the extent to which they agree (strongly disagree, somewhat disagree, somewhat agree, strongly agree) with statements describing their knowledge, emotional, and social self-worth. One WPASWI item from each of the self-worth domains was chosen for the pilot phase. Based upon results of the pilot phase, the EMA survey was modified for the test phase and two items were chosen to assess each domain, for a total of six items from the WPASWI. Examples include: "RIGHT NOW - My knowledge about physical activity affects the way I feel about myself." (knowledge self-worth) "RIGHT NOW - I feel it is important to take time to be physically active today." (emotional self-worth) "RIGHT NOW - I need to know I have friends or family to support my commitment to exercise in order to feel good about myself." (social self-worth)

Two items from the Physical Self-Perception Profile (Fox & Corbin, 1989) will be used to measure perceived body attractiveness and physical condition, both important subdomains of physical self-worth. Women will be asked the extent to which they agree (strongly disagree, somewhat disagree, somewhat agree, strongly agree) with the following statements:

"RIGHT NOW - I feel confident about the appearance of my body." (body attractiveness) "RIGHT NOW - I am confident in my level of physical conditioning and fitness." (physical condition)

In summary, the EMA survey used in the test phase of this study will include eleven items assessing momentary activity (1) (Dunton et al., 2012); self-efficacy (1) (McAuley, 1993), general self-worth (1) (Messer & Harter, 1986); knowledge (2), emotional (2), and social (2) self-worth (Huberty et al., 2013); and physical self-worth (2) (Fox & Corbin, 1989).

Women will also be asked to wear a GENEActiv accelerometer for the duration of their participation in the study (14 days for the pilot phase and 28 days for the test phase). All participants will receive their GENEActiv during the initial intake appointment and will return the device during a schedule appointment with a researcher. Women not local to the Phoenix area will receive and return their GENEActiv by mail. As part of wearing the activity monitor, women will also be asked to log their wear time, wake time, and bedtime. All participants will receive comprehensive feedback on their time spent in sedentary, light, moderate, and vigorous activity each day.

During the intake appointment, women will also be asked to complete the full-length questionnaires upon which the EMA survey was developed (i.e., Exercise Self-Efficacy Scale [McAuley, 1993], Adult Self-Perception Profile [Messer & Harter, 1986], WPASWI [Huberty et al., 2013], Physical Self-Perception Profile [Fox & Corbin, 1989]), a demographics questionnaire, and a regular PA questionnaire (Past-Week Modifiable Activity Questionnaire [Gabriel et al., 2010]).

ELIGIBILITY:
Inclusion Criteria:

* 35-64 years of age
* English speaking
* Able to ambulate
* Own a mobile phone with access to text messaging and cellular Internet
* Able to receive text messages from a short code
* Agree that user rates will apply when receiving text messages and completing assessments

Exclusion Criteria:

* Males
* Not within age range; children
* Non-English speaking
* Unable to ambulate
* Do not own a mobile phone with access to text messaging or cellular Internet
* Not able to receive text messages from a short code
* Do not agree to accept user rates

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nationally recruited sample of active and inactive middle-aged women (35-64 years-old)
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Self-Worth | 28 days
  General self-worth: One item from the general self-worth subscale of the Adult Self-Perception Profile (Messer & Harter, 1986) Knowledge, emotional, and social self-worth: Six items (two per self-worth domain) from the Women's Physical Activity Self-Worth Inventory (Huberty et al., 2013) Physical self-worth: Two items from the Physical Self-Perception Profile (Fox & Corbin, 1989)
Physical Activity - Accelerometer | 28 days
  GENEActiv wrist-worn accelerometer

SECONDARY OUTCOMES:
Exercise Self-Efficacy | 28 days
  One item from the Exercise Self-Efficacy Scale (McAuley, 1993)
Current Activity | 28 days
  One item from a recent EMA study by Dunton et al. (2012)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — Arizona State Unversity

REFERENCES:
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] White SM, Wojcicki TR, McAuley E. Social cognitive influences on physical activity behavior in middle-aged and older adults. J Gerontol B Psychol Sci Soc Sci. 2012 Jan;67(1):18-26. doi: 10.1093/geronb/gbr064. Epub 2011 Jul 9. PMID 21743038
- [Background] Huberty JL, Ransdell LB, Sidman C, Flohr JA, Shultz B, Grosshans O, Durrant L. Explaining long-term exercise adherence in women who complete a structured exercise program. Res Q Exerc Sport. 2008 Sep;79(3):374-84. doi: 10.1080/02701367.2008.10599501. PMID 18816949
- [Background] Segar ML, Eccles JS, Richardson CR. Type of physical activity goal influences participation in healthy midlife women. Womens Health Issues. 2008 Jul-Aug;18(4):281-91. doi: 10.1016/j.whi.2008.02.003. Epub 2008 May 12. PMID 18468920
- [Background] Pettee Gabriel K, McClain JJ, Schmid KK, Storti KL, Ainsworth BE. Reliability and convergent validity of the past-week Modifiable Activity Questionnaire. Public Health Nutr. 2011 Mar;14(3):435-42. doi: 10.1017/S1368980010002612. Epub 2010 Sep 15. PMID 20843404
- [Background] McAuley E. Self-efficacy and the maintenance of exercise participation in older adults. J Behav Med. 1993 Feb;16(1):103-13. doi: 10.1007/BF00844757. PMID 8433355
- [Background] Dunton GF, Liao Y, Kawabata K, Intille S. Momentary assessment of adults' physical activity and sedentary behavior: feasibility and validity. Front Psychol. 2012 Jul 30;3:260. doi: 10.3389/fpsyg.2012.00260. eCollection 2012. PMID 22866046
- [Background] Esliger DW, Rowlands AV, Hurst TL, Catt M, Murray P, Eston RG. Validation of the GENEA Accelerometer. Med Sci Sports Exerc. 2011 Jun;43(6):1085-93. doi: 10.1249/MSS.0b013e31820513be. PMID 21088628
- [Background] Huberty J, Vener J, Gao Y, Matthews JL, Ransdell L, Elavsky S. Developing an instrument to measure physical activity related self-worth in women: Rasch analysis of the Women's Physical Activity Self-Worth Inventory (WPASWI). Psychology of Sport and Exercise 14(1): 111-121, 2013.
- [Background] Messer BJ, Harter S. Manual for the adult self-perception profile. University of Denver, 1986.
- [Background] Fox KR, Corbin CB. The physical self-perception profile: Development and preliminary validation. Journal of Sport and Exercise Psychology 11: 408-430, 1989.
- [Derived] Ehlers DK, Huberty J, Buman M, Hooker S, Todd M, de Vreede GJ. A Novel Inexpensive Use of Smartphone Technology for Ecological Momentary Assessment in Middle-Aged Women. J Phys Act Health. 2016 Mar;13(3):262-8. doi: 10.1123/jpah.2015-0059. Epub 2015 Aug 13. PMID 26284689